CLINICAL TRIAL: NCT06175481
Title: Correlation Between Popliteal Vein Compliance and Venous Clinical Severity Score
Status: Completed | Type: Observational
Sponsor: Hao Liu (Other)
Responsible Party: Sponsor-Investigator, Hao Liu, Clinical Professor, Guangdong Second Provincial General Hospital
Organization: Guangdong Second Provincial General Hospital (Other)
Other Study IDs: HaoLiu
Record Dates: First submitted 2023-11-28; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-10

CONDITIONS: Chronic Venous Disease (CVD), Vein Compliance, Venous Clinical Severity Score (VCSS)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
  Interventions: Other: Popliteal Vein Compliance
- experimental group
  Interventions: Other: Popliteal Vein Compliance

INTERVENTIONS:
Other: Popliteal Vein Compliance — Compliance of the popliteal vein is calculated as the distensibility, with the ratio of functional caliber/native caliber/cuff pressure value ( mmHg-1 ).

SUMMARY:
When the liquid flow increases, the luminal caliber's stretching amplitude decreases, leading to a higher hydraulic pressure according to Poiseuille's law. In this study, investigators measured the caliber change of the popliteal vein under a rated pressure gradient and evaluated the relationship between popliteal vein compliance and venous clinical severity score (VCSS).

ELIGIBILITY:
Inclusion Criteria:

* C1 to C6 disease using the CEAP (clinical, etiologic, anatomic, pathophysiologic) classification.

Exclusion Criteria:

* acute or chronic thrombosis of deep veins, previously received intravenous surgery or injection sclerotherapy, ankle brachial index<0.90, and concomitant cardiovascular, pulmonary, renal, or metabolic diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were prospectively enrolled in Guangdong Second Provincial General Hospital from May 2023 to October 2023. All participants gave their voluntary consent.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Compliance of the popliteal vein | May 2023 to October 2023
  Compliance of the popliteal vein is calculated as the distensibility, with the ratio of functional caliber/native caliber/cuff pressure value

CONTACTS AND LOCATIONS:
Locations (1):
- Hao Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu H, Li L, Wei W, Tang Y, Liu L, Xiao C. Correlation between popliteal vein functional diameter and the severity of chronic venous disease. Phlebology. 2025 Jul;40(6):415-419. doi: 10.1177/02683555241310531. Epub 2024 Dec 21. PMID 39708049